CLINICAL TRIAL: NCT06295575
Title: The Effect of Probiotics on Intestinal Barrier Function and Intestinal Flora in Infants With Congenital Heart Disease Undergoing Cardiopulmonary Bypass
Brief Title: Effect of Probiotics on Patients With Congenital Heart Disease Following Cardiopulmonary Bypass
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing Children's Hospital (Other)
Responsible Party: Principal Investigator, Zhixuan Zhang, Principal investigator, Nanjing Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZZhang
Record Dates: First submitted 2024-02-21; First posted 2024-03-06 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-02

CONDITIONS: Congenital Heart Disease; Intestinal Disease; Dysbiosis
MeSH Terms: conditions — Heart Defects, Congenital; Intestinal Diseases; Dysbiosis | interventions — Lacteol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Active Comparator): In treatment group, patients received 1×109 colony forming units (CFU) /day of probiotic, which was provided by Hangzhou Grand Biologic Pharmaceutical INC (Zhejiang, China) in the form of freeze-dried powder containing Bifidobacterium infantis and Lactobacillus with a density of 109 CFU/g. The probiotic powder was mixed with lactose and portioned into sachets with the help of Nanjing Medical University Central Pharmacy.
  Interventions: Dietary Supplement: probiotics containing Bifidobacterium infantis and Lactobacillus
- Control group (Placebo Comparator): Patients in the control group received lactose as placebo. The placebo was packed in sachets and provided in the same way as treatment group.
  Interventions: Dietary Supplement: placebos containing lactose

INTERVENTIONS:
Dietary Supplement: probiotics containing Bifidobacterium infantis and Lactobacillus — Patients were provided with probiotics containing Bifidobacterium infantis and Lactobacillus. This intervention was started the day after patients' administration and lasted until the day before discharge.
  Arms: Treatment group
Dietary Supplement: placebos containing lactose — Patients received lactose as placebo.This intervention was started the day after patients' administration and lasted until the day before discharge.
  Arms: Control group

SUMMARY:
A randomized, controlled study including infants with non-cyanosis congenital heart disease (CHD) in need of surgical correction involving cardiopulmonary bypass (CPB) was established. Infants aged 1 month to 1 years were enrolled between June 2021 and July 2022. The patients in treatment group were supplied with probiotics consisting of Bifidobacterium infantis and Lactobacillus perioperatively and patients in control group were provided with placebo. Data concerning patients' clinical outcome such as diarrhea were collected. Blood samples were collected for measurement of fatty acid binding protein 2 (FABP2), diamine oxidase (DAO), d-lactic acid (D-LA) and C-reactive protein (CRP). Stool samples were collected to investigate the changes of intestinal flora.

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis of CHD requiring surgical repair with the use of CPB
* age greater than 37 weeks corrected gestational age and less than 1 year old

Exclusion Criteria:

* Patients with inherited metabolic disease, history of intestinal surgery, preexisting gastrointestinal pathology (such as NEC, IBS, inflammatory bowel disease, chronic intestinal obstruction or diarrhea), immunity dysfunction or received antibiotics, probiotics or hormone-replacement therapy within 2 months before enrollment were excluded from the study

Ages: 1 Month to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
incidence of morbidity | up to 1 months
  morbidity of intestinal diseases including pathology verified by imageological examination such as necrotizing enterocolitis (NEC) and acute intestinal obstruction or bowel dysfunction such as diarrhea
gastrointestinal functional recovery indicators | up to 1 months
  starting time of full enteral feeding (hours post-surgery) and duration of gastrointestinal decompression were recorded for assessment of gastrointestinal functional recovery
biomarkers | after anesthesia induction preoperatively and at 24 hour postoperatively
  serum concentrations of biomarkers of intestinal barrier function and intestinal inflammation, namely IFABP, DAO, D-LA and CRP, were recorded
microbiome | before surgery: within 24 hours after enrollment in the control group and within 24 hours preoperatively in the treatment group after surgery:between 48 and 72 hours in both groups
  16s rDNA sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Zhixuan Zhang, Principal Investigator — Nanjing Children's Hospital; Xiaoxu Liu, Study Director — Department of Cardiothoracic Surgery, Children's Hospital of Nanjing Medical University, Nanjing, Jiangsu Province, China
Locations (1):
- Children's Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
Data collation and website construction have not yet been completed